CLINICAL TRIAL: NCT04084158
Title: A Phase II, Randomized, Open Label, Multi-center Design Study of Toripalimab Given Before and After Concurrent Chemoradiotherapy in Patients With Locally Advanced Esophageal Squamous Cell Carcinoma
Brief Title: A Study of Toripalimab Combined With Concurrent Chemoradiotherapy for Locally Advanced Esophageal Squamous Cell Carcinoma.
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: combination arm delevelped significant poor prognosis
Sponsor: Zhejiang Cancer Hospital (Other)
Collaborators: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IESO001
Record Dates: First submitted 2019-09-05; First posted 2019-09-10 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: Esophageal Squamous Cell Carcinoma; PD-1 antibody
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — toripalimab; Albumin-Bound Paclitaxel; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Toripalimab+chemoradiation (Experimental): Induction immunotherapy: Toripalimab injection (JS001) 3mg/kg IV q 14 days x 2 cycles.
  Concurrent Chemoradiotherapy: Starting within 4 weeks after the first cycle induction immunotherapy. carboplatin AUC = 2 + albumin-bound paclitaxel 60 mg/m2 or paclitaxel liposome 45 mg/m2 or paclitaxel 45 mg/m2 IV weekly x 6 weeks concurrent with radiation to a total dose of 50.4 Gy given in 1.8 Gy fractions daily x 28 fractions.
  Progression of disease (PD): The progress of the disease will be assessed within 4 weeks after concurrent chemoradiotherapy. Patients without disease progression continue to receive consolidation and adjuvant therapy.
  Consolidation chemotherapy: carboplatin AUC = 6 + albumin-bound paclitaxel 260 mg/m2 or paclitaxel liposome 135 mg/m2 or paclitaxel 135 mg/m2 IV q 21 days x 6 cycles.
  Adjuvant immunotherapy:Toripalimab injection (JS001) 3mg/kg IV q 14 days up to 1 year.
  Interventions: Drug: Toripalimab injection (JS001); Drug: Paclitaxel, Albumin-Bound; Radiation: Radiotherapy; Drug: Platinum-Based Drug
- chemoradiation (Active Comparator): Concurrent Chemoradiotherapy: carboplatin AUC = 2 + albumin-bound paclitaxel 60 mg/m2 or Liposome paclitaxel 45 mg/m2 or paclitaxel 45 mg/m2 IV weekly x 6 weeks concurrent with radiation to a total dose of 50.4 Gy given in 1.8 Gy fractions daily x 28 fractions.
  Progression of disease (PD): The progress of the disease will be assessed within 4 weeks after concurrent chemoradiotherapy. Patients without disease progression continue to receive consolidation therapy.
  Consolidation chemotherapy: carboplatin AUC = 6 + albumin-bound paclitaxel 260 mg/m2 or paclitaxel liposome 135 mg/m2 or paclitaxel 135 mg/m2 IV q 21 days x 6 cycles.
  Interventions: Drug: Paclitaxel, Albumin-Bound; Radiation: Radiotherapy; Drug: Platinum-Based Drug

INTERVENTIONS:
Drug: Toripalimab injection (JS001) — Toripalimab injection (JS001) is a humanized IgG4 monoclonal antibody against the programmed death-1 (PD-1) receptor, blocks the interaction of PD-1 with its ligands and promotes T cell activation in preclinical studies.
  Arms: Toripalimab+chemoradiation
Drug: Paclitaxel, Albumin-Bound — Paclitaxel
Radiation: Radiotherapy — PTV 50.4Gy/28 fractions, PGTV 61.6Gy/28 fractions, once a day, 5 days a week.
Drug: Platinum-Based Drug — carboplatin

SUMMARY:
The purpose of this study is to explore the efficacy and safety of Toripalimab injection (JS001) given before and after concurrent chemoradiotherapy for locally advanced esophageal squamous cell carcinoma.

DETAILED DESCRIPTION:
This was a randomized, open label and multi-center phase II clinical study, which aimed to evaluate the efficacy and safety of Toripalimab injection (JS001) induction immunotherapy, plus concurrent chemoradiation, and successive Toripalimab injection (JS001) maintenance immunotherapy relative to those of standardized concurrent chemoradiation for locally advanced esophageal squamous carcinoma patients that could not receive surgical treatment or refuse surgery. All patients conforming to the inclusion and exclusion criteria were assigned as the experimental arm and control arm at the ratio of 1:1 through the stratified block randomization method. Prior to concurrent chemoradiation, the experimental arm was given anti-PD-1 antibody Toripalimab injection (JS001) for 2 cycles, concurrent chemoradiation was initiated within 4 weeks after the induction immunotherapy, then patients were evaluated within 4 weeks after the completion of concurrent chemoradiation. Those who had not achieved PD were given 2 cycles of consolidation chemotherapy, and Toripalimab injection (JS001) was continued to at most 1 year or to identified disease progression, intolerable toxicity, or the subjects asked to withdraw initiatively, or researchers judged that the subjects should withdraw from the study. The control arm was given concurrent chemoradiation alone, with sequential consolidation chemotherapy for 2 cycles. The primary endpoint is progression-free survival (PFS), Secondary end points include objective response rate (ORR), overall survival (OS), duration of response (DoR), time to distant metastasis (TTDM).

ELIGIBILITY:
Inclusion Criteria:

1. 18≤age≤75.
2. Histologically or cytologically confirmed esophageal squamous carcinoma.
3. Patients must have unresectable disease as assessed by thoracic surgeons or refuse surgical treatment.
4. The investigator confirmed at least one measurable lesion according to RECIST 1.1.
5. Stage II-IVA (AJCC 8th)
6. No adjacent organs infringed confirmed by endoscopic ultrasonography (T1-3).
7. ECOG PS 0-1.
8. FEV1>0.8L
9. Life expectancy is not less than 12 weeks.
10. No prior chemotherapy, radiotherapy, biotherapy, immunotherapy or other anti-tumor treatment for esophageal cancer.
11. Adequate organ function defined at baseline as: 1) ANC ≥1.5×109 /L，PLt ≥100×109 /L，Hb ≥90 g/L; 2) TBIL ≤1.5×ULN, ALT ≤2.5ULN, AST ≤2.5ULN, BUN and Cr ≤1×ULN or Ccr ≥50ml/min (Cockcroft-Gault formula); 3) INR ≤1.5×ULN or PT ≤1.5×ULN (If the patient is receiving anticoagulant therapy, PT should be within the intended use range of the anticoagulant drug); 4) Myocardial zymogram is within normal range.
12. Women of childbearing age must have taken reliable contraceptive measures or have a pregnancy test (serum or urine) within 7 days prior to enrollment and the results are negative. Besides, subjects should agree to use effective methods of contraception during the trial and within 2 months of the last dose of anti-PD-1 antibody. For male subjects whose spouse are of childbearing age, effective contraceptive methods should be used during the trial and within 2 months after the last dose of anti-PD-1 antibodies;
13. Subject volunteers to join the study, Signs informed consent, has good compliance and can cooperate with follow-up.

Exclusion Criteria:

1. Those with prior or concurrent uncured malignant tumor. cured skin basal cell carcinoma, cervical cancer and superficial bladder cancer were excluded.
2. Esophageal cancer patients with primary multifocal lesions.
3. Those with the pathology of small cell esophageal carcinoma, esophageal adenocarcinoma or mixed carcinoma.
4. Primary esophageal squamous carcinoma with active hemorrhage of the primary lesion within 2 months.
5. Those with primary esophageal lesion that was closely related to tracheal bronchus and great vessels, and were evaluated with a great risk of perforation and massive bleeding by the researchers.
6. Patients with any active autoimmune disease or autoimmune disease history (such as interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, myocarditis, nephritis, hyperthyroidism, and hypothyroidism (those with normal thyroid function after hormone replacement therapy could be enrolled); those with leucoderma or childhood asthma that was completely relieved and required no intervention during adulthood could be enrolled, while asthma patients requiring bronchodilators and medical intervention should not be enrolled.
7. Patients with uncontrolled cardiovascular disease: grade II and above myocardial ischemia or myocardial infarction, and poorly-controlled arrhythmia (including the QTc interval of ≥470 ms); those with grade III-IV cardiac insufficiency according to the NYHA criteria, or those whose echocardiography revealed left ventricular ejection fraction (LVEF) of <50%; and those having myocardial infarction within 1 year.
8. Those with active infection or fever of >38.5 ℃ with unknown cause during the screening period and before the first administration (patients with tumor-induced fever judged by the researchers could be enrolled).
9. Those with interstitial lung disease or active non-infectious pneumonia history or evidence.
10. Those with congenital or acquired immunodeficiency (such as those with HIV infection), active hepatitis B (HBV-DNA≥104 copies/ml) or hepatitis C (positive hepatitis C antibody, and the HCR-RNA was higher than the lower limit of detection of the analysis method).
11. Those who had previously received other PD-1 antibody treatment or PD-1/PD-L1 targeted immune therapy.
12. Those who were known to be allergic to paclitaxel, carboplatin, macromolecular protein preparation, or any anti-PD-1 antibody component.
13. Subjects who required to use corticosteroids (prednison dose of > 10 mg/day) or other immunosuppressors for systemic treatment within the first 7 days of research. In the absence of active autoimmune disease, glucocorticoids at physiological dose (≤ 10 mg/day prednison or equivalent drug), inhalation or local application of steroid and adrenocortical hormone replacement treatment with prednison at the dose of > 10 mg/day.
14. Those receiving anti-tumor monoclonal antibody (mAb) and targeted small molecule treatment within 4 weeks before the initial use of the research drug, or those with unrecovered adverse events induced by the previous treatment (namely, grade ≤ 1 or reaching the baseline level). Apart from subjects with ≤ grade 2 nervous lesion or ≤ grade 2 alopecia, any subject that had received major surgery should sufficiently recover from the toxic reaction and/or complication resulted from the surgical intervention before the initiation of treatment.
15. Those who were within 4 weeks before the initial use of the research drug (subjects that had entered the follow-up period were calculated at the final use of experimental drug or instrument) or those who were participating other clinical research.
16. Patients should be inoculated with live vaccine within 4 weeks before the initial use of research drug, inactivated viral vaccine specific to seasonal influenza for injection was allowed, but the nasal use of live attenuated influenza vaccine was not allowed.
17. Pregnant women or breast-feeding women.
18. Subjects who had other factors that might force them to terminate the research ahead of time, such as the development of other severe disease (including mental disease) that required combined treatment, seriously abnormal laboratory examination value, and family or social factors that might affect the subject safety or experimental data collection, as judged by the researchers.

    -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-09-07 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
PFS | 2 years
  Progression-Free Survival

SECONDARY OUTCOMES:
Objective Response Rate | analysis is completed 4 weeks after concurrent chemoradiation
  Ratio of CR and PR (RECIST 1.1) in all subjects
OS | 3 years
  Overall Survival
DoR | 2 years
  Duration of Response
TTDM | 3 years
  Time to distant Metastasis

CONTACTS AND LOCATIONS:
Overall Officials: Chen Ming, MD, Principal Investigator — Zhejiang Cancer Hospital; Yujin Xu, MD, Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No